CLINICAL TRIAL: NCT01153412
Title: Effect of Osteopathic Manipulation on Postural Stability in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, Rita Patterson, PhD, Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-087
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Balance Control in Elderly
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Control group no intervention
- Osteopathic Manipulative Treatment (Experimental): Osteopathic Manipulative medicine group
  Interventions: Other: Osteopathic Manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — Osteopathic manipulation to determine balance and stability in elderly
  Arms: Osteopathic Manipulative Treatment

SUMMARY:
Postural stability and balance are defined as the body's ability to return the body back to its equilibrium point when exposed to a perturbation. This exploratory project is based on the hypotheses that decreased balance (increased sway as measured by the center of pressure of the body during quiet standing) causes an increased risk of falls and osteopathic manipulative treatment can improve postural balance. To test these hypotheses, the investigators will investigate the kinematics (study of the way the body moves) of postural balance in two cohorts of healthy elders, those receiving manipulation and those not receiving manipulation. We hypothesize that OMT is effective to increase postural stability, balance.

DETAILED DESCRIPTION:
Postural stability and balance are defined as the body's ability to return the body back to its equilibrium point when exposed to a perturbation. This exploratory project is based on the hypotheses that decreased balance(increased sway as measured by the center of pressure of the body during quiet standing) causes an increased risk of falls and osteopathic manipulative treatment can improve postural balance. To test these ideas, the investigators will investigate the kinematics(study of the way the body moves)of postural balance in two cohorts of healthy elders, those receiving manipulation and those not receiving manipulation. We hypothesize that OMT is effective to increase postural stability, balance.

Specific Aims Aim 1: To measure balance in a cohort of healthy elders(age 65 and over)using a force plate to measure center of pressure in the Anterior/posterior and medial-lateral directions during quiet standing with the eyes open, with the eyes closed and during a Romberg test.

Aim 2: To evaluate the effectiveness of OMT to improve balance in a healthy elderly population. We will observe the progression of improvement in balance in one group who will receive OMT for four weeks compared to the other who will not receive OMT.

Aim 3: To examine any potential impact and efficacy of OMT on cardiac and circulatory responses by measuring blood flow and circulation.

ELIGIBILITY:
Inclusion Criteria:

* 65 years ofage and older
* Healthy
* Male and Female

Exclusion Criteria:

* Self report of a condition that could impair balance, such as otoneurologic, musculoskeletal or neurological diseases.
* Under the age of 65

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Balance | 30 seconds
  Center of Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rita Patterson, PhD, Principal Investigator — UNTHSC

IPD SHARING:
Plan to Share IPD: Yes
Can provide de-identified center of pressure data from the project.

REFERENCES:
- [Result] Lopez D, King HH, Knebl JA, Kosmopoulos V, Collins D, Patterson RM. Effects of comprehensive osteopathic manipulative treatment on balance in elderly patients: a pilot study. J Am Osteopath Assoc. 2011 Jun;111(6):382-8. doi: 10.7556/jaoa.2011.111.6.382. PMID 21771924